CLINICAL TRIAL: NCT05290779
Title: Ultrasound Versus Fluoroscopy-guided Selective Lumbar Nerve Root Injection for Treatment of Radicular Pain
Brief Title: Ultrasound Versus Fluoroscopy-guided Selective Lumbar Nerve Root Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Islam Ahmed Bakr Mohammed, Director, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: US vs. FL SNRB injection
Record Dates: First submitted 2022-02-25; First posted 2022-03-22 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Lumbar Radiculopathy
Keywords: lumbar radicular pain; selective nerve root injection; ultrasound selective lumbar nerve root injection
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ultrasound (Active Comparator): selective lumbar nerve root steroid injection under ultrasound guidance.
  Interventions: Procedure: selective lumbar nerve root injection
- fluoroscopy (Sham Comparator): selective lumbar nerve root steroid injection under fluoroscopy guidance.
  Interventions: Procedure: selective lumbar nerve root injection

INTERVENTIONS:
Procedure: selective lumbar nerve root injection — selective lumbar nerve root steroid injection for treatment of radicular pain.

SUMMARY:
The study is conducted to compare pain relief, accuracy and safety and radiation exposure of selective lumbar nerve root injection for lumbar radicular pain using ultrasound guidance versus fluoroscopy guidance

DETAILED DESCRIPTION:
Radicular pain is believed to be induced by irritation or inflammation of a nerve root caused by mechanical pressure or chemical irritation from degeneration herniation or rupture of intervertebral disc .Nerve root steroid injection is the most commonly performed minimally invasive technique for treatment of radicular pain in lumbar spine.The mechanism of action of steroids is to reduce inflammation by reduction in proinflammatory mediators around the nerve root, causing reduction in pain levels . Although Fluoroscopy guided technique is the most widely accepted method in lumbar selective nerve root injection, but recently ultrasound technique has gained acceptance among physicians due its reliability, efficacy, real-time guidance of injection and reduction of radiation exposure. Real-time guidance of injection provided by ultrasonography allows for good identification of the spinous process and adjacent structures such as lamina, zygapophyseal articulations and transverse process allowing for safer and potentially equally effective injection technique. The patients are randomly allocated into two groups; one group will receive injection under fluoroscopy guidance and the other group will receive injection under ultrasound guidance. The two groups are compared in terms of pain relief, accuracy and safety and radiation exposure.

ELIGIBILITY:
Inclusion Criteria:

* adult patients aged 18-60 years .
* Both sexes .
* With unilateral chronic lumbar radicular pain for more than 3 months.
* Cooperative and oriented patients.
* All patients are diagnosed by a neurologist for radicular low back pain through clinical presentation, medical examinations, computed tomography (CT), or magnetic resonance imaging (MRI).

Exclusion Criteria:

* Uncontrolled diabetes.
* Infection at the site of injection.
* Spine fractures.
* Previous back surgery.
* Progressive neurologic disorders.
* Fever.
* Peripheral neuropathy.
* Presence of motor or sphencteric disturbance.
* Bilateral radicular pain.
* Allergy to substance of injection.
* Patients with body mass index (BMI) more than 35.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2022-04-12 (Actual); Study Completion 2022-05-16 (Actual)

PRIMARY OUTCOMES:
improvement of visual analogue score of pain | 3 months
  evaluation of pain relief using visual analogue score on a scale from 0 to 10 with higher scores mean worse outcome
improvement of Oswestry disability index score for back pain | 3 months
  evaluation of pain relief using Oswestry disability index score on a scale from 0% to 100% with the higher scores mean worse outcome.

SECONDARY OUTCOMES:
safety of technique | 3 months
  comparing rate of complications
radiation exposure | 1 hour
  time of x-ray radiation exposure during procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Amany K Abu Elhusein, PhD, Study Chair — Professor of Anesthesia and intensive care, MiniaU.; Abd ELraheem M Mohamed, MD, Study Director — Assistant professor of Anesthesia and intensive care, AsuitU..
Locations (1):
- Faculty of medicine, Minya, Egypt